CLINICAL TRIAL: NCT07270445
Title: Effect of Virtual Reality Use on Preoperative Anxiety: A Prospective, Randomized, Controlled Interventional Study (VeRA-Study)
Brief Title: Effect of Virtual Reality Use on Preoperative Anxiety
Acronym: VeRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vera Guttenthaler (Other)
Responsible Party: Sponsor-Investigator, Vera Guttenthaler, Clinical Study Coordinator, University of Bonn
Organization: University of Bonn (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-291-BO
Record Dates: First submitted 2025-11-17; First posted 2025-12-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anxiety
Keywords: VR glasses; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality glasses (Experimental)
  Interventions: Device: Virtual reality glasses
- Control (No Intervention)

INTERVENTIONS:
Device: Virtual reality glasses — he VR headset creates an immersive environment that allows patients to distance themselves from the real surroundings. Calming visual and auditory stimuli can be presented through the VR headset, promoting relaxation. Initial results have shown that this application can reduce preoperative anxiety and postoperative pain perception in adult patients and may offer a non-pharmacological alternative to benzodiazepines and opioids. The Effect of Virtual Reality on Preoperative Anxiety: A Meta-Analysis of Randomized Controlled Trials by Chiu demonstrated a reduction in anxiety in the intervention group among adults, with an effect size of 0.57.
  Arms: Virtual reality glasses

SUMMARY:
The aim of this study is to investigate the effect of a non-pharmacological intervention-the use of a virtual reality headset-on preoperative anxiety levels in patients. For this purpose, both psychometric instruments (STOA and APAIS questionnaires) and objective physiological and EEG parameters are used. Patients who do not receive any additional intervention will form the control group.

The study was designed as a prospective, randomized, controlled, interventional study at the University Hospital Bonn. Patients aged 18 years and older who are scheduled to undergo elective surgery and who have no visual, hearing, or language impairments will be included in the study.

The primary objective of the study is the reduction of preoperative anxiety. The hypothesis is that preoperative use of the VR headset reduces perioperative anxiety, stress, and pain.

DETAILED DESCRIPTION:
The investigators are planning a prospective, randomized controlled study with the aim of reducing patients' preoperative anxiety through VR use and improving postoperative pain and anxiety levels. After obtaining informed consent, patients will be randomly assigned to either the control or the intervention group. Stratification will be performed based on the presence of relatives during the preoperative process (yes/no) to ensure an even distribution of this potential confounding factor.

Patient anxiety will be assessed using the State-Trait Operation Anxiety (STOA) and the Amsterdam Preoperative Anxiety and Information Scale (APAIS) questionnaires. Stress and pain will be measured using the Numeric Rating Scale (NRS) from 0 to 10. A baseline assessment of simulator sickness will be performed using the Simulator Sickness Questionnaire (SSQ), which evaluates three symptom groups: nausea, oculomotor discomfort, and disorientation.

Following the questionnaires, patients will undergo EEG monitoring using the BIS device (Bispectral Index Monitor). The BIS is a medical monitoring device widely used in anesthesiology to measure anesthesia depth based on EEG data. Different mental states are associated with specific EEG frequency bands (alpha, beta, gamma, delta, and theta), and EEG is a well-established method for evaluating emotions. Alpha waves are linked to increased relaxation and reduced sympathetic arousal, and enhancing alpha waves in neurofeedback therapy has been shown to reduce anxiety. Beta waves are often associated with motor tasks and cognitive processing, and studies have also shown that increased beta activity correlates with higher anxiety levels. Anxiety affects beta activity by shifting power from lower to higher frequencies. All this suggests that a decrease in alpha-beta ratios (ABR) and low-high beta ratios (BR) may indicate the presence of stress and anxiety. EEG monitoring will continue until the first postoperative hour. Continuous EEG recording allows intraoperative and postoperative EEG patterns to be correlated with anxiety scores and postoperative pain.

During the preoperative process, all patients will be monitored for blood pressure, respiratory rate, oxygen saturation, and heart rate. These measurements will be used to objectively document the effects of sympathetic nervous system activation due to anxiety.

The control group will receive routine clinical care, while the intervention group will undergo a 20-minute VR session. During the session, patients will watch videos of natural landscapes and listen to calming music and nature sounds through headphones to promote relaxation. If any discomfort occurs, the session will be immediately stopped. At the end of the VR session, the SSQ will be repeated. Before entering the operating room, anxiety, stress, and pain levels will be assessed again.

During the first postoperative hour, anxiety, stress, pain, and patient satisfaction with the study procedure will be evaluated. Satisfaction with the study and the VR intervention will be measured using the NRS and a satisfaction questionnaire specific to the VR session. Patients will also be assessed for delirium using the Nursing Delirium Screening Scale (Nu-DESC). Throughout the entire process, all patients will be continuously monitored using EEG/BIS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent
* All consecutive patients undergoing elective, outpatient, or inpatient surgery
* No communication difficulties (e.g., hearing impairment) and good command of the German language
* No visual impairment
* Planned extubation immediately after surgery

Exclusion Criteria:

* Patients undergoing emergency surgery
* Patients with documented psychiatric disorders (e.g., bipolar disorder), confusion, or epilepsy
* Individuals admitted due to a court or official order
* Expected non-compliance with the study protocol
* Expected admission to an intermediate care unit (IMC) or intensive care unit (ICU)
* Patients receiving sedative or anxiolytic medication for premedication
* Patients with pacemakers or defibrillators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The change of anxiety | From date of randomization until the date of first documented progression, assessed up to 8 hours
  The STOA evaluates anxiety on two levels: the long-term, personality-related tendency toward surgical anxiety (trait) and the current state of anxiety (state), with cognitive and affective components. The STOA-State scale includes 10 items rated on a 4-point scale from 0 ("Not at all") to 3 ("Very much"), yielding a total score of 0-30. The STOA-Trait scale includes 20 items rated from 0 ("Almost never") to 3 ("Almost always"), with a total score of 0-60.
The change of anxiety | From date of randomization until the date of first documented progression, assessed up to 8 hours
  The APAIS is a validated, brief instrument with 20 items, assessing anxiety related to anesthesia and the surgical procedure. Anxiety scores range from 4 (no anxiety) to 20 (high anxiety), and the total score ranges from 6 to 30.

SECONDARY OUTCOMES:
Change of preoperative stress and pain | From date of randomization until the date of first documented progression, assessed up to 8 hours
  The Numeric Rating Scale (NRS) is a measurement tool in which participants indicate the intensity of their stress or pain on a scale from 0 to 10. A score of 0 represents "no stress/pain," while a score of 10 represents "very severe stress/pain."
Delirium incidence in the recovery room | From date of randomization until the date of first documented progression, assessed up to 8 hours
  The NuDESC is a brief, validated tool used to screen for delirium in hospitalized patients. It assesses five key domains: disorientation, inappropriate behavior, inappropriate communication, hallucinations, and psychomotor retardation. Each item is scored from 0 to 2, where 0 indicates "absent," 1 indicates "mild," and 2 indicates "severe." The total score ranges from 0 to 10, with higher scores reflecting greater severity of delirium.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bonn, Bonn, Germany